CLINICAL TRIAL: NCT04072042
Title: A Biomarker Driven, Open Label, Phase II Study of VEGFR2 Inhibitor Apatinib in Patients With Recurrent or Refractory Advanced Bone and Soft Tissue Sarcoma
Brief Title: BIOmarker Driven Trial of VEGFR2 Inhibitor in Advanced or Metastatic Sarcoma
Acronym: BIOVAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weibin Zhang, MD, PhD., Director of the orthopaedics department, Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2019LLS167
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: In each of the treatment arm, we recruit patients according to the biomarker status and hypothesize that the anti-angiogenic therapeutic efficay would be higher than historical control as a biomarker-driven approach.
Who Masked: Outcomes Assessor
Masking Description: Radiological Assessment of tumor will be independently reviewed by outcome assessor, who is blinded to patient biomarker status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VEGFR SNP-Positive Sarcoma Arm (VEGFR-AtoG) (Experimental): In this arm, patients with VEGFR2-604 A>G single nucleotide polymorphism (SNP) were recruited for the efficacy analysis.
  Biomarker positive patients will receive Apatinib 250mg tablet by mouth, bid. Biomarker negative patients are treated with the same regimens as a non-comparative, non-randomized, pragmatic control without a pre-specified sample size.
  Interventions: Drug: Apatinib monotherapy
- CSF1-Positive Sarcoma Arm (CSF1-high) (Experimental): In this arm, patients with CSF1-positivity were recruited for the efficacy analysis. CSF1-positivity is defined as CSF1 copy number amplification and/or CSF1 expression ≥ 30% by immunohistochemistry (IHC) in the sarcoma tumor specimen according to the institutional pathological review.
  Biomarker positive patients will receive Apatinib 250mg tablet by mouth, bid. Biomarker negative patients are treated with the same regimens as a non-comparative, non-randomized, pragmatic control without a pre-specified sample size.
  Interventions: Drug: Apatinib monotherapy
- 4q12 amplicon-Positive Sarcoma Arm (4q12-amp) (Experimental): In this arm, patients with 4q12 amplicon (4q12-amp) were recruited for the efficacy analysis. 4q12-amp is defined as copy number amplification of chromosome segment 4q12 detected by fluorescence in situ hybridization (FISH) in the sarcoma tumor specimen according to the institutional pathological review.
  Biomarker positive patients will receive Apatinib 250mg tablet by mouth, bid. Biomarker negative patients are treated with the same regimens as a non-comparative, non-randomized, pragmatic control without a pre-specified sample size.
  Interventions: Drug: Apatinib monotherapy

INTERVENTIONS:
Drug: Apatinib monotherapy — patients will receive Apatinib 250mg tablet by mouth, bid.
  Other Names: VEGFR inhibitor; Rivoceranib

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Apatinib monotherapy for relapsed or refractory advanced bone and soft tissue sarcoma with VEGFR-2 (KDR) 604A>G polymorphism as predictive biomarker

DETAILED DESCRIPTION:
After standard chemotherapy and surgery for the localized disease, pulmonary metastases of bone and soft tissue sarcoma occurs in up to 40% of cases and still remain challenging without satisfactory regimen. Apatinib has been reported as a novel oral kinase inhibitor of receptor tyrosine (TKI) targeting VEGFR2 as an angiogenesis inhibitor. Previous studies indicated that Apatinib, as well as other novel VEGFR inhibitor (such as Regorafenib, Cabozantinib, Pazopanib ), showed a promising anti-sarcoma activity with a 4 month progression free rate (PFR) ranging from 40 to 60% in advanced bone and soft tissue sarcoma after multi-line chemotherapy failure. However, the significant inter-individual variability of the agents suggests a lack of predictive biomarker for its clinical use. Furthermore, up to 10~30% of patients may encounter pneumothorax, a potentially life-threatening consequence. Other common debilitating adverse effects (AEs) include surgical wound complication, hand foot skin reaction, etc.

Our preliminary data (Presented in ESMO poster session and ESMO Asia oral session in 2019) suggests that rs2071559_VEGFR2 604A>G polymorphism is associated pulmonary tumor cavitation (predisposes one to pneumothorax), hair depigmentation, superior anti-tumor efficacy. Therefore, the investigators aim to explore the clinical signficance of pneumothorax incidence as well as the efficacy of Apatinib monotherapy for advanced bone and soft tissue sarcoma in association with VEGFR-2 (KDR) 604 genotype. We aim to further conduct our clinical study in two cohorts: the observational study cohort and the prospective clinical trial cohort.

In the observational cohort, we recruited patients with anti-angiogenic TKIs who encounter pneumothorax during the course of the treatment from nation-wide as a real world study. We review the radiological features of their tumor (such as cavitation, location, etc.) and the medical history of the pre-treatment. We then prospectively follow up the oncological outcomes and the respiratory outcomes given that all pneumothoraces are treated with multidisciplinary approaches to minimize the adverse effect of pneumothoax and maximize the duration of response to anti-angiogenic TKIs. We expect that the patients with pneumothorax (an efficacy related toxicity), if managed actively, will have a durable progression-free survival compared to historical control. Blood samples will also be collected for genotyping VEGFR2 604A>G polymorphism status as a validation to our preliminary findings.

In the prospective clinical trial cohort, we formally designed a prospective single-arm, open-label, biomarker-driven phase II clinical trial to explore the efficacy of Apatinib, a novel anti-angiogenic oral inhibitor, in biomarker-based selective patients as follows: With all comers(biomarker positive and negative) allowed to be enrolled, only VEGFR-2 (KDR) 604A>G polymorphism positive will be measured for the primary endpoint of the study according to our sample size estimation . The primary objective is to hypothesize that the progression-free rate (PFR) of Apatinib in this population is ≥ 70% at 4 months (tremendous higher than non-biomarker driven historical control), against the null hypothesis of PFR ≤ 50% as in the general sarcoma patients. Using Simon's two stage design, we are going to recruit 9 biomarker-positive patients in the first stage. If the primary objective was reached in >3 patients, study continue to recruit a total of 28 biomarker-positive patients. The primary endpoint will be considered met if 18 or more patients achieve PFR at 4 months. Considering the potential lost to follow-up, a total of 30 patients with biomarker positive is needed in this trial. Biomarker-negative patients will be analyzed as a non-comparative control without pre-specified sample size, which is expected to be similar to the historical control of advanced bone and soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. age between 8 and 65 years;
2. diagnosis of histologically confirmed advanced bone and soft tissue sarcoma excluding adipocytic tumor;
3. identification of pulmonary lesion is mandatory;
4. refractory to prior treatment consisted of standard National Comprehensive Cancer Network (NCCN) guideline recommended first-line chemotherapy;
5. Eastern Cooperative Oncology Group(ECOG) performance status 0-2 with a life expectancy >3 months;
6. adequate renal, hepatic, and hemopoietic function;normal or controlled blood pressure;
7. advanced stage that complete surgical resection of all lesions are infeasible;
8. no serious thoracic comorbidities with adequate pulmonary function for daily living;
9. previously treated with tyrosine kinase inhibitors (TKIs) for less than 8 weeks but off treatment due to manageable complications such as wound complications or pneumothorax without adequate interventions. The complications is resolved and disappeared at enrollment.

Exclusion Criteria:

1. have had other kinds of malignant tumors at the same time;
2. cardiac insufficiency or arrhythmia;
3. uncontrolled complications, such as diabetes mellitus and so on;
4. coagulation disorders or Hemorrhagic diseases ;
5. pleural or peritoneal effusion that needs to be handled by surgical treatment;
6. combined with other infections or wound complications;
7. wound dystrophy, poor soft-tissue around implantation risky of non-healing given angiogenesis inhibitor at baseline;
8. previously treated with VEGFR TKIs for more than 8 weeks
9. previous treated with VEGFR TKIs but off treatment due to oncological assessment or dose-limiting complications given adequate interventions.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
4 month-progression free rate (PFR) in each of the 3 cohorts | 4 months from recruitment
  Each arm of the study is analyzed separately with the progression free rate (PFR) as the primary outome measure. PFR is defined as the proportion of patients that are progression-free according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
progression free rate (PFR) in biomarker negative control in each of the 3 cohorts | 4 months from recruitment
  The proportion of patients with negative biomarker that are progression-free according to RECIST 1.1
progression free survival(PFS) between biomarker positive and negative patients in each of the 3 cohorts | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  The difference of PFS between biomarker positive and biomarker negative control with log-rank test in each of the 3 cohorts
Correlation of biomarker positivity with overall survival (OS) | Baseline until death, assessed for an average of 24 months
  Correlation of biomarker positivity with OS to RECIST 1.1 among all comers in each of the 3 cohorts
ORR, DCR and DOR between biomarker positive and negative patients in each of the 3 cohorts | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  The difference of objective response rate (ORR), disease control rate (DCR) and durable of response (DOR) between biomarker positive and biomarker negative patients according to RECIST 1.1 in each of the 3 cohorts
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 8 months
  The occurrence of each adverse events(AEs), severe AEs(SAEs) and death according the CTCAE_5.0
Correlation of KDR polymorphism with pulmonary lesion cavitation/pneumothorax | 4 months from recruitment
  Correlation of KDR 604 AA，AG，GG genotype with the incidence of pulmonary lesion cavitation or pneumothorax among all comers in cohort 1 (VEGFR2-AtoG cohort)
Correlation of KDR polymorphism with hair depigmentation | 4 months from recruitment
  Correlation of KDR 604 AA，AG，GG genotype with the incidence of hair depigmentation among all comers in cohort 1 (VEGFR2-AtoG cohort)
Correlation of CSF1R polymorphism (rs10079250) with wound complication | through study completion, an average of 8 months
  Correlation of CSF1R (rs10079250) genotype with the incidence of wound complications among all comers
Correlation of PDGFRα polymorphism (rs35597368) with hand foot skin reaction | through study completion, an average of 8 months
  Correlation of PDGFRα (rs35597368) genotype with the incidence of hand foot skin reaction among all comers
Early identification of AEs as predictive biomarker | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  to correlate the incidence of targeted therapy related AEs （pulmonary lesion cavitation, pneumothorax, hair depigmentation) with the PFS

OTHER OUTCOMES:
Exploratory outcome: Subgroup analysis of progression-free survival(PFS) | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  The PFS for each subgroups in terms of clinicopathological characteristics (age, gender, histological type, solitary or multiple metastases, unilateral or bilateral metastases, early or late metastases, calcifying or non-calcifying lesions, with or without lesion cavitation, with or without AEs [especially pneumothorax, hand-foot skin reactions, hair depigmentation], etc
Exploratory outcome: the molecular analysis of tumor sample in each of the 3 cohorts | through study completion, an average of 8 months
  To explore the molecular basis underlying the difference of biomarker positive and negative sub-cohorts using next generation sequencing
Exploratory outcome: the pattern of disease progression between different cohorts and different sub-group within each cohort | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  to compare the growth pattern/ distribution of pulmonary versus extrapulmonary lesion at baseline and at disease progression between different cohorts and different sub-group within each cohort
Exploratory outcome: 1.0-mm CT scan for pulmonary assessment | Baseline until disease progression or death, whichever occurs first, assessed for an average of 8 months
  to compare the diagnostic value of the 1.0 mm versus 5.0 mm CT scan for the radiological evaluation of small lung nodule as tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Zhang, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China